CLINICAL TRIAL: NCT02270112
Title: Enhanced Diagnostics for Early Detection of Atrial Fibrillation - DETECT AF Trial
Brief Title: Enhanced Diagnostics for Early Detection of Atrial Fibrillation
Acronym: DETECT-AF
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Jens Eckstein, MD, PhD, University Hospital, Basel, Switzerland
Other Study IDs: EKNZ:2014-080
Record Dates: First submitted 2014-10-03; First posted 2014-10-21 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial electrophysiology; stroke; vascular stiffness
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paroxysmal Af: No Intervention is planned. All patients receive a 5 Minute ECG and have their pulse recordes by an iPhone.
  Interventions: Device: ECG

INTERVENTIONS:
Device: ECG — Patients receive a 5 Minute ECG recording and have their pulse recorded by an iPhone.

SUMMARY:
Paroxysmal atrial fibrillation can only be diagnosed during episodes when the arrhythmia is present.

The investigators hypothesize that the activation of the atrial myocardium resulting in the p-wave of the ecg should display abnormalities in diseased atria which are vulnerable for AF.

DETAILED DESCRIPTION:
In the first part of this trial different diagnostic techniques to detect arrythmogenic substrates of atrial fibrillation will be tested. If suitable parameters can be identified, a follow up trial to identify patients at risk for AF will be conducted before a stroke happens.

Parameters tested are

1. Electrophysiological differences between patients with paroxysmal AF and no history of AF
2. "Vascular Stiffness" detected by an iPhone app

All patients will undergo a cardiogoniometrie and a pulse wave analysis with an iPhone. Each exam takes 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation in sinus rhythm at presentation

Exclusion Criteria:

* acute cerebral trauma
* antiarrhythmic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All inhospital and outpatient patients of our Institution with known paroxysmal AF are screened for eligebility. Control Group is equally recruted from patients of our intitution matching the studygroup.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Beat to beat variation of the electrical activation vector of the atrium | Once during the exam (baseline) - No further follow up planned
  Test if the beat to beat Variation of the electrical activation of the atrium differentiates between the group of patients with paroxysmal AF and no AF in history.

SECONDARY OUTCOMES:
Averaged slope of pressure-curve | Once during exam (5min, baseline) - No further follow up planned
  Test if the steepness of the slope of the pressure curve recorded with the iPhone differs between the two Groups.
Averaged slope of pressure-curve | Once during exam (5min, baseline) - No further follow up planned
  Test if the steepness of the slope of the pressure curve recorded with the iPhone correlates with cardiovascular risk factors.
Heart rate variability | Once during exam (5min, baseline) - No further follow up planned
  Test if heart rate variability recorded with the iPhone differs between the two Groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, MD, PhD, Principal Investigator — Universityhospital Basel
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Brasier N, Engelter S, Kolbitsch T, Tabord A, Knobeloch J, Kuhne M, Conen D, Traenka C, Kreutzberger T, Vollmin G, Eckstein J. The quest for indicators of paroxysmal atrial fibrillation in sinus rhythm - the DETECT AF trial. Acta Cardiol. 2019 Aug;74(4):301-307. doi: 10.1080/00015385.2018.1493248. Epub 2018 Aug 19. PMID 30122130